CLINICAL TRIAL: NCT06463704
Title: General Pre-Trial Screening Protocol for Enrollment of Volunteers Into Infectious Diseases Research Protocols
Brief Title: General Pre-Trial Screening Protocol for Infectious Diseases Research
Status: Recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Kathryn Stephenson, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2023P000266
Record Dates: First submitted 2024-05-23; First posted 2024-06-18 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational cohort for potential study volunteers: This is a general screening protocol to develop a registry of potential volunteers for our clinical trials. There is no intervention to be administered.
  Interventions: Other: There is no intervention

INTERVENTIONS:
Other: There is no intervention — There is no intervention

SUMMARY:
The purpose of this general screening protocol is to facilitate recruitment into studies conducted at the Center for Virology and Vaccine Research (CVVR) or Division of Infectious Diseases at Beth Israel Deaconess Medical Center. This general screening protocol will help to determine the eligibility of potential volunteers for any vaccine or therapeutic trials open for recruitment or soon to be opened.

DETAILED DESCRIPTION:
The purpose of this general screening protocol is to facilitate recruitment into studies conducted at the Center for Virology and Vaccine Research (CVVR) and Division of Infectious Diseases at Beth Israel Deaconess Medical Center. This protocol will help us to determine whether a volunteer is eligible for completing the screening process and which protocols might best be suited to the participant.

Volunteers will be adults interested in participating in a clinical trial, such as a vaccine or therapeutic study, and particularly for studies conducted as part of the HIV Vaccine Trials Network. Occasionally, the screening protocol may be used for an observational study. This general screening protocol will help to determine the eligibility of potential volunteers for any clinical trials open for recruitment or soon to be opened. No investigational products will be administered under this protocol. All main vaccine or intervention studies will be submitted as separate applications to the appropriate regulatory agency as required by the sponsor.

Prescreening of volunteers may be done via telephone using an already approved script and RedCap questionnaire. Following the prescreening, the volunteer will be scheduled for an in-person clinic visit with a study clinician (MD, NP or RN). All participants in this study will be screened for safety, including a physical exam, vital signs and laboratory testing. This is to ensure that participants meet the appropriate inclusion and exclusion criteria related to safety in a clinical trial. The following study procedures will be performed at the Clinical Research Center at BIDMC:

1. Informed Consent process completed before any other study activities are conducted
2. Demographics
3. Medical history
4. Review of current medications
5. Targeted physical exam including vital signs
6. Behavioral risk assessment to determine risk of acquiring HIV
7. Contraception status
8. Blood or urine collection: on average, most safety screening laboratory tests will require no more than 60mL of blood which will be resulted in BIDMC's clinical laboratory. A urine sample may be collected for people of childbearing potential to determine pregnancy status.

Laboratory tests will be checked against eligibility criteria of open or soon-to-be opened clinical trials. If a test or exam result suggest that further medical evaluation or treatment may be necessary, the participant will be notified and referred to their care provider for further treatment. A copy of test results will be provided if requested.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at time of consent
* Available to participate for the planned duration of the clinical trials for which screening is being done
* Capable of giving signed informed consent

Exclusion Criteria:

• A condition, based on clinical judgement, which requires active medical intervention or monitoring to avert serious danger to the participant's health or well-being

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Volunteers will be adults interested in participating in a clinical trial, such as a vaccine or therapeutic study, and particularly for studies conducted as part of the HIV Vaccine Trials Network.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2034-06 (Estimated)

PRIMARY OUTCOMES:
Distribution of demographic variables | At enrollment
  Race, ethnicity, gender and sex at birth
Number of participants who subsequently enroll in another study | From date of enrollment until the date of enrollment in a subsequent study or up to 52 weeks, whichever comes first
  The number of participants in the general screening protocol who go on to enroll in another study

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided